CLINICAL TRIAL: NCT05600660
Title: Orelabrutinib, Rituximab and Methotrexate (OR-MTX) in Newly Diagnosed Primary Central Nervous System Lymphoma: a Single Arm, Multicenter, Phase 2 Study
Brief Title: Orelabrutinib,Rituximab and Methotrexate in Newly Diagnosed Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0407
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary Central Nervous System Lymphoma; Orelabrutinib; Methotrexate; Lenalidomide
MeSH Terms: interventions — orelabrutinib; Rituximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OR-MTX (Experimental): Experimental arm will be treated with OR-MTX regimen(Orelabrutinib plus Rituximab and Methotrexate) for 6 cycles as initiate induction. After 6 cycles of induction chemotherapy, autologous Hematopoietic Stem Cell Transplantation (AHSCT) will be performed for transplantation eligible patients . Thereafter, Orelabrutinib maintenance chemotherapy will be given up to one year. Follow-ups should be taken up to the first 2 years. The primary endpoint is objective response rate (ORR) and secondary endpoint includes Progression free survival (PFS), overall survival (OS), and adverse events.
  Interventions: Drug: Orelabrutinib; Drug: Rituximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Orelabrutinib — Orelabrutinib will be given as 150 mg/d orally 72h after MTX infusion or MTX clearance, every 21 days for 6 cycles during induction treatment.
  Daily Orelabrutinb will be administered as maintenance treatment for up to 1 year or until disease progression, intolerable toxicity, death, informed consent withdrawal or lost of follow up (whichever occurs first).
Drug: Rituximab — 375mg/m2 intravenous infusion d1, every 3 weeks for 1 cycle, 6 cycles will be prescribed for induction therapy.
Drug: Methotrexate — 3.5g/m2 intravenous infusion for 4 hours in d1, every 21 days for 1 cycle, 6 cycles will be prescribed.

SUMMARY:
It is a single arm, multicenter, phase 2 study to explore the efficacy and safety study of OR-MTX chemotherapy（Orelabrutinib, Rituximab and Methotrexate）as first-line regimens in the treatment of newly diagnosed primary central nervous system lymphoma. Objective response rate is the primary endpoint.

DETAILED DESCRIPTION:
This is a single arm, multicenter, phase 2 study designed to evaluate the efficacy and safety of Orelabrutinib, rituximab and methotrexate as first-line regimens in the treatment of newly primary central nervous system lymphoma. A total of 28 patients plan to participate in this study to receive a total 6 cycles of induction chemotherapy followed by Orelabrutinib maintenance chemotherapy up to one year. After 6 cycles of induction chemotherapy, autologous Hematopoietic Stem Cell Transplantation (AHSCT) will be performed for transplantation eligible patients . Follow-ups should be taken up to the first 2 years. The primary endpoint is objective response rate (ORR) and secondary endpoint includes Progression free survival (PFS), overall survival (OS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Primary Central Nervous System (CNS) lymphoma Age range 18-75 years old.
2. Eastern Cooperative Oncology Group performance status 0 to 3.
3. Previously untreated. Patients treated with steroid alone are eligible.
4. Measurable disease was defined as at least ≥1.0cm in short-diameter by MRI.
5. Life expectancy of ≥ 3 months (in the opinion of the investigator).
6. Participants must be able to understand and be willing to sign a written informed consent document.
7. Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 6 months after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 6 months after the last dose.

   Women of childbearing potential must have a negative plasma pregnancy test upon study entry.
8. Adequate renal function: Estimated glomerular filtration rate (GFR) or estimated creatinine clearance (CrCl) ≥ 50 mL/min;Serum creatinine ≤ 2 times the upper limit of normal.
9. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value & Bilirubin < 2 X upper normal value.
10. Adequate hematological function: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL.
11. Must be able to tolerate lumbar puncture and MRI/CT.
12. Ability to swallow oral medications.

Exclusion Criteria:

1. Patient with systemic, non-CNS lymphoma metastatic to the CNS.
2. Patient is concurrently using other approved or investigational antineoplastic agents.
3. Presence of active hepatitis B virus(HBV) infection (HBsAg positive and HBV-DNA≥ 104), hepatitis C virus(HCV) infection, acquired and congenital immunodeficiency diseases include but not limited to HIV.
4. Patient is allergic to components of the study drug.
5. Patient has an active concurrent malignancy requiring active therapy.
6. Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, uncontrolled congestive heart failure, uncontrolled hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening.
7. Patient is known to have an uncontrolled active systemic infection.
8. Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk.
9. Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive plasma human chorionic gonadotropin(hCG) laboratory test of > 5 mIU/mL.
10. The patient is unwell or unable to participate in all required study evaluations and procedures.
11. Drug abuse, medical, psychological or social conditions which may interfering with subjects' participation in the study or evaluation of the results.
12. History of intracranial hemorrhage or clinically significant stroke within 6 months prior to first day of study treatment
13. History of significant gastrointestinal disease that would limit absorption of oral medications.
14. Warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Use of low molecular weight heparin and novel oral anticoagulants (eg. rivaroxaban, apixaban) is permitted if required.
15. Concurrent use of a moderate or strong inhibitor or inducer of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers prior to starting the study drug.
16. Known bleeding diathesis (e.g. von Willebrand's disease), hemophilia, or active bleeding.
17. History of invasive fungal infection, including invasive aspergillosis, or known active tuberculosis.
18. Patients considered unsuitable to participate in the study by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | At the end of Cycle 6 chemotheray (each cycle is 21 days)
  The objective response rate is defined as the proportion of patients with a response of complete response(CR) or partial response(PR).

SECONDARY OUTCOMES:
Progression free survival | 2years
  From date of patients sign informed consent until the date of progression or death or the date of last follow-up time, whichever came first, assessed up to 2 years
Treatment-related adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
ctDNA mutation and mean ctDNA concentration in serum and cerebrospinal fluid | Baseline, every two months for up to 2 years after treatment
  Types of ctDNA mutations and frequency are measured by next generation sequencing. The mean ctDNA concentration is the concentration of ctDNA expressed as mean tumor molecules /ml at specific time points.
The levels of cytokine concentration in serum and cerebrospinal fluid | Baseline, every two months for up to 2 years after treatment
  The levels of cytokine will be analyzed by ELISA in all patients recruited. The cytokine profile includes IL-6, IL-10, TNF-α, IFN-γ, IL-2 and IL-4

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Xiao XB, Weng YQ, Jiang HW, Li X, Xie J, Bao CQ, Qian WB. Orelabrutinib combined with rituximab and high-dose methotrexate as induction therapy in newly diagnosed primary central nervous system lymphoma. Invest New Drugs. 2025 Jun;43(3):679-686. doi: 10.1007/s10637-025-01548-1. Epub 2025 May 27. PMID 40425940